CLINICAL TRIAL: NCT02931214
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GMI-1359 in Healthy Adult Subjects
Brief Title: Placebo-Controlled Single Dose Study to Evaluate Safety and Pharmacokinetics of GMI-1359 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMI-1359-101
Record Dates: First submitted 2016-09-06; First posted 2016-10-12 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Healthy Subjects; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GMI-1359 (Experimental): Dose escalation
  Interventions: Drug: GMI-1359
- Placebo (Experimental): Dose escalation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GMI-1359
  Arms: GMI-1359
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate safety and pharmacokinetics of single ascending IV doses of GMI-1359 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending IV dose study conducted at one study center in the United States. Safety will be assessed throughout the study and serial blood samples and urine samples will be collected for the safety and pharmacokinetic assessment of GMI-1359.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or females, 19-60 years of age (inclusive).
2. Medically healthy with no clinically significant screening results.
3. Females of childbearing potential must either be sexually inactive (abstinent) for 3 months prior to dosing or be using an acceptable birth control method
4. Females must have a negative pregnancy test at the time of screening and prior to dosing for inclusion in the study.
5. Understands the study procedures in the informed consent form, and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated.
2. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subjects by their participation in the study.
3. Normal clinical laboratory values.
4. Normal heart rate and blood pressure.
5. Blood donation or significant blood loss within 56 days prior to dosing.
6. Plasma donation within 7 days prior to dosing.
7. Participation in another clinical trial within 28 days prior to dosing.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse events | 15 days
  Treatment related adverse events as a measure of safety and tolerability of GMI-1359

SECONDARY OUTCOMES:
Pharmacokinetics | 48 hours
  Cmax (peak plasma concentration)
Pharmacokinetics | 48 hours
  AUC (area under the curve)
Pharmacokinetics | 48 hours
  Tmax (time to peak plasma concentration)
Pharmacodynamics | 48 hours
  CD34 cell measurement

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No